CLINICAL TRIAL: NCT05513755
Title: Randomized Trial of Cardioneuroablation in Reflex Syncope Treatment (CARDIOSYE Trial)
Brief Title: Cardioneuroablation in Reflex Syncope (CARDIOSYRE Trial)
Acronym: CARDIOSYE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación de investigación HM (Other)
Collaborators: Hospital HM Monteprincipe (Unknown); Fundacion Dexeus (Other); Hospital de Basurto (Other); Hospital Universitario La Paz (Other); Hospital Clínico Universitario de Valladolid (Other); Hospital Universitario Marqués de Valdecilla (Other); Hospital Vall d'Hebron (Other); Hospital Clinic of Barcelona (Other); Hospital General Universitario de Alicante (Other); Hospital Clinico Universitario San Cecilio (Other); University Hospital Virgen de las Nieves (Other); Puerta de Hierro University Hospital (Other); Hospital San Pedro de Alcantara (Other); Hospital of Navarra (Other); Complejo Hospitalario Universitario de Albacete (Other); Hospital Universitario Ramon y Cajal (Other); Complejo Hospitalario Universitario de Badajoz (Other)
Responsible Party: Principal Investigator, Teresa Barrio, principal investigator, Fundación de investigación HM
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cardioneuroablation in Syncope
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Reflex Syncope
Keywords: reflex syncope; cardioneuroablation; randomized
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardioneuroablation (Experimental)
  Interventions: Procedure: cardioneuroablation
- Conventional treatment (counter-pressurre maneuver, drugs or pacemaker) (No Intervention)

INTERVENTIONS:
Procedure: cardioneuroablation — Endocardical radiofrequency ablation of vagal ganglia located close to pulmonary veins antra and interatrial septum.
  Arms: Cardioneuroablation

SUMMARY:
Background: Reflex syncope is a disease of benign etiology but in severe cases it can be disabling and it carries a risk of severe trauma. Today, there is no proven etiological treatment and only palliative treatments are used, namely a change in hygienic and dietary habits, certain drugs or, in the most severe cases, the implantation of a pacemaker. Cardioneuroablation is a novel technique that acts by ablating the parasympathetic ganglia located on the external walls of the atria. Several prospective series with promising results have been published, but there are no randomized studies that have validated its efficacy compared to conventional treatment.

Methods: The CARDIOSYRE study is a multicenter, randomized, single-blinded study of patients with reflex syncope. The aim is to recruit, between June 2022 and June 2025, 92 patients with reflex cardioinhibitory syncope in 15 centers and randomize them (1:1 ratio) to two treatment groups: 1) cardioneuroablation intervention; 2) conventional treatment (control group). The primary end-point will be the time to the first syncope and the secondary end-point will be the total incidence of syncope after one year of follow-up. At least 20 recurrences of syncope are expected during a 1-year follow-up. A relative risk of 0.3 and a statistical power of 80% are assumed. The follow-up will be carried out at 3, 6 and 12 months. Cox models will be used to estimate adjusted Hazard ratios.

ELIGIBILITY:
Inclusion Criteria:

* Patients with reflex syncope (two or more episodes in the last year) and cardioinhibitory response (documentation of asystole >3 seconds coinciding with syncope or >6 seconds outside of syncope or cardioinhibitory response on the tilt test) defined such as heart rate < 40 bpm for at least 10 seconds or asystolic pause > 3 seconds

Exclusion Criteria:

* Patients under 18 years
* Any pathology or medical condition that limits survival to less than one year;
* Illegal drug use, chronic alcoholism, or total alcohol use >80 g/d
* Participation in a clinical trial conducted with drugs or use of a drug in an experimental state during the year prior to inclusion
* Patients institutionalized for chronic treatment, with a lack of autonomy and with the impossibility of carrying out clinical follow-ups
* Patients with pacemakers, patients with intrinsic disease of the cardiac conduction system or bundle branch block
* Patients with structural heart disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
time to the first syncope | 12 months
  time from the randomization to the first syncope

SECONDARY OUTCOMES:
number of syncopes during the follow-up period | 12 months
  number of syncopes during the follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- Teresa Barrio Lopez, Madrid, Spain